CLINICAL TRIAL: NCT04797884
Title: A Randomized Study of Intrabucally Administered Electromagnetic Fields Versus Placebo for Patients With Child-Pugh A or B With Advanced Hepatocellular Carcinoma
Brief Title: Electromagnetic Fields Versus Placebo For Child-Pugh A and B Patients With Advanced Hepatocellular Carcinoma
Acronym: ARTEMIS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: THERABIONIC INC. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00072592; 20231793 (Other: WCG IRB); R44CA256984 (NIH)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Child-Pugh A and B
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TheraBionic Arm - Active Arm (Experimental): For subjects who are randomized to the active arm, the device will be programmed with hepatocellular carcinoma-specific modulation frequencies and will be activated for >200 one-hour treatment sessions.
  Interventions: Device: TheraBionic Device; Device: Quality of Life Assessment
- Placebo Arm (Placebo Comparator): For subjects randomized to the placebo arm, the device will not emit any hepatocellular carcinoma-specific modulation frequencies and will be activated for >200 one-hour treatment sessions.
  Interventions: Device: Placebo Device; Device: Quality of Life Assessment

INTERVENTIONS:
Device: TheraBionic Device — Each treatment day consists of three courses of 60-minute treatments to be administered in the morning, at noon, and in the evening. Each 6-week treatment period will be considered a cycle of treatment. With the exception of the first 60-minute treatment, which will be delivered at one of the recruiting site, all other treatments will be self-administered at the patient's home.
  Arms: TheraBionic Arm - Active Arm
Device: Placebo Device — Each treatment day consists of three courses of 60-minute treatments to be administered in the morning, at noon, and in the evening. Each 6-week treatment period will be considered a cycle of treatment. With the exception of the first 60-minute treatment, which will be delivered at the recruiting site, all other treatments will be self-administered at the patient's home.
  Arms: Placebo Arm
Device: Quality of Life Assessment — Ancillary services

SUMMARY:
The primary goals of this study are to compare overall survival and quality of life in subjects with Child-Pugh A or B advanced hepatocellular carcinoma when treated with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

DETAILED DESCRIPTION:
Primary Objectives

To compare the overall survival between subjects with advanced hepatocellular carcinoma treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

To compare the patient-reported disease-related symptoms between subjects with advanced hepatocellular carcinoma treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

Secondary Objectives

To compare progression-free survival between subjects treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

To compare safety and tolerability between subjects treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

To compare the effect on levels of alpha-fetoprotein between subjects treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

To compare global treatment side effect bother between subjects treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

To compare patient-rated symptomatic adverse events between subjects treated either with a device emitting radiofrequencies modulated at specific frequencies or with a device emitting unmodulated radiofrequencies.

ELIGIBILITY:
Inclusion Criteria:

Biopsy-proven HCC that is locally advanced or metastatic OR

* Patients without biopsy confirmation are also eligible if they meet one of the following criteria:

  1. Radiologic diagnosis of HCC as per the AASLD guidelines OR
  2. Liver cirrhosis AND a liver mass that shows arterial phase hyperenhancement on triphasic computed tomography (CT) or MRI, AND either:

     * Is ≥ 20 mm with either non-peripheral portal washout or an enhancing capsule OR
     * Is 10-19 mm with non-peripheral portal venous washout AND an enhancing capsule
* For Child-Pugh A participants: treatment failure (defined as documented radiological progression) and/or intolerance to at least two prior treatments with approved or experimental systemic therapies including atezolizumab plus bevacizumab, sorafenib, lenvatinib, regorafenib, cabozantinib, ramucirumab, nivolumab, nivolumab plus ipilimumab, pembrolizumab or any other approved or experimental first line and/or second line therapy.
* Child-Pugh B participants are not required to have received any prior treatment.
* Measurable disease according to RECIST v 1.1.
* At least one target lesion that has not previously received any local therapy, such as surgery, radiation therapy, hepatic arterial embolization, transarterial chemoembolization (TACE), hepatic arterial infusion, radio-frequency ablation, percutaneous ethanol injection or cryoablation, unless it has subsequently progressed by 20% or more according to RECIST v 1.1 and mRECIST for HCC.
* Patients with Child-Pugh A or B (at time of enrollment) as defined by the parameters contained in the Child-Pugh Calculator. Subjects with Child-Pugh score of B8-B9 may be included if they have:

  * Albumin ≥ 2.8 mg/l AND
  * Total Bilirubin ≤ 3.0mg/l.
* ECOG performance status of 0-2.
* At least 2 weeks must have elapsed since administration of any anticancer treatment prior to initiation of protocol therapy.
* Patients must be greater than or equal to 18 years old and must be able to understand and sign an informed consent.
* Female patients of childbearing potential and their partners and male patients must agree to use adequate contraception during the period of study treatment.

Exclusion Criteria:

* Known leptomeningeal disease. (Previously treated, asymptomatic central nervous system (CNS) metastases are eligible).
* Fibrolamellar HCC or combined hepatocellular-cholangiocarcinoma (cHCC-CC).
* Prior treatment with the TheraBionic Device.
* Patients with any of the following within the 12 months prior to registration: uncontrolled/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism.
* Pregnant or breastfeeding women.
* Patients with another active malignancy within the past one year except for treated cervical cancer in situ, treated in situ carcinoma of the bladder or treated non-melanoma carcinoma of the skin, low-risk prostate cancer not requiring active treatment, treated T1/T2 glottic cancer, treated stage 0 or stage I breast cancer not requiring adjuvant therapy or treated non-invasive bladder cancer.
* Patients receiving calcium channel blockers and any agent blocking L-type of T-type Voltage Gated Calcium Channels, e.g., amlodipine, nifedipine, ethosuximide, ascorbic acid (vitamin C), etc. unless their medical treatment is modified to exclude calcium channel blockers prior to enrollment.
* Patients with curative treatment options available, including surgery or radiofrequency ablation, as assessed by their physician.
* Patients receiving other anticancer treatments.
* Patients that do not agree to be followed according to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Baseline to 6 months
  Overall survival assessment will be recorded in days and will represent the period starting at the date of treatment initiation and finishing at the date of patient death. Living patients at the time of analysis will have the date of last contact (consultation visit or phone contact) used to define overall survival.
Quality of Life Survey | Baseline to 6 months
  Patient-reported hepatobiliary-specific disease-related symptoms will be assessed by the 18-item FACT-Hepatobiliary (Hep) subscale every cycle for the first 6 cycles then every other cycle thereafter, at the end of treatment, and at every 3 months during follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 2 years
  Progression free survival (PFS) will be compared between groups using a 2-sided log rank test. Kaplan-Meier survival curves for PFS will also be generated and median progression free survival and corresponding 95% confidence intervals will be estimated for each group
Proportion of Patients With Disease Control | At 4 months and 6 months and up to 2 years
  Proportion of patients who respond and the corresponding 95% Clopper Pearson exact confidence intervals. Patients who are removed from study before the 6-month time point will be considered to not have disease control at that time point.
Proportion of Participants That Are Progression Free | At 12 weeks, 4 months and 6 months and up to 2 years
  we will determine the proportion of patients who are progression free after 12 weeks (after 2nd 6-week visit) and compare this between groups using a Fisher's exact test. In addition, the corresponding 95% Clopper Pearson exact confidence intervals will be calculated for the 4 month and 6 month progression free survival rates.
Incidences of Adverse Events - CTCAE version 5.0 | Up to 28 days after study treatment administration or until death
  Using Common Terminology Criteria for Adverse Events [CTCAE], version 5.0, type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities will be assessed.
Changes in Alfa-Fetoprotein Levels | 6 months
  Investigators will examine whether these is any association between the AFP levels (potential biomarker for response) and the objective response observed for each participant. Average alfa-fetoprotein levels will be examined over time, and these changes in alfa-fetoprotein rates after 6 months will be examined for each Response category (complete response/ partial response/ stable disease/ progressive disease) and tested using a 1-way ANOVA to see if the change in AFP level differs by response category.
Functional Assessment of Cancer Therapy-General (FACT-G) Item GP5 | At baseline and every 6 weeks up to 6 months
  Participants will answer a single item question from the FACT-G questionnaire "I am bothered by side effects of treatment" Scoring scale of 0 (not at all) to 4 (very much) to assess for side effects to assess for patient rated treatment tolerability.
Frequency of Adverse Events - PRO-CTCAE | At baseline and every 8 weeks up to 6 months
  The frequency and nature of patient-reported symptomatic adverse events will be assessed using 10 items from the PRO-CTCAE item library. PRO-CTCAE items will assess mucositis (2 items; severity, interference), dry mouth (1 item, severity), fatigue (2 items; severity, interference), decreased appetite (2 items; severity, interference), nausea (1 item, severity), and headache (2 items; severity, interference) to measure potential adverse events associated with the study intervention. Participants will select the one response that best describes their experience with a scoring scale(s) of None to Very Severe or Not at all to Very Much.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie K Pasche, MD, Principal Investigator — THERABIONIC INC.
Locations (7):
- United States (7):
  - Tampa General Hospital, Tampa General Cancer Center, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Knight Cancer Institute, Portland, Oregon
  - Thomas Jefferson University Hospital, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - DHR Health Advanced Care Center, DHR Oncology Institute, Edinburg, Texas
  - University of Texas Health Science Center, Mays Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators of this project will make the non-proprietary results and accomplishments of the research plan available to the research community and to the public at large by the timely release and sharing of data. As a means of sharing knowledge, the investigators supported by this grant will seek to publish the original research in primary scientific journals. The investigators will also assert copyright in scientific and technical articles based on data produced under the grant where necessary. For each publication that results from the grant-supported research, we will include an acknowledgment of NIH grant support and follow guidelines regarding free access to published materials. Information on each publication resulting from work performed under the NIH grant supported project will be included in the annual and/or final progress report submitted to the NIH awarding office.
  Proprietary developments will be protected using intellectual property rights.
Supporting Information: Study Protocol, SAP
Time Frame: Within six months of data publication